CLINICAL TRIAL: NCT02988076
Title: A Prospective, Double Blind, Randomized, Controlled, Multisite Study to Evaluate the Utility, Safety, and Efficacy of Using PEER Interactive to Inform Medication Prescription to Subjects With a Primary Diagnosis of a Depressive Disorder(SMART-MD)
Brief Title: Study to Evaluate the Safety and Efficacy of PEER Interactive to Inform Medication Prescription for Subjects With a Primary Diagnosis of Depression
Acronym: SMART-MD
Status: Suspended | Phase: Phase 2 / Phase 3 | Type: Interventional
Why Stopped: Lack of recruiting at primary study site
Sponsor: MYnd Analytics (Industry)
Collaborators: Mount Sinai Hospital, New York (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CNSR012
Record Dates: First submitted 2016-12-07; First posted 2016-12-09 (Estimated); Last update posted 2020-07-30 (Actual); Status verified 2020-07

CONDITIONS: Depression
Keywords: database; probability; response; depression; medication; quantitative; electroencephalogram
MeSH Terms: conditions — Depression

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Masking Description: The subject is masked as to assignment to Control or Treatment Group. The subject acts as the blinded rater - providing the primary outcome measure - the Quick Inventory of Depressive Symptomatology - 16 Item Self report
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control (No Intervention): The Control group subjects will undergo all procedures e.g. medication washout and baseline electroencephalogram, administered to the Treatment/Experimental group. A clinician treating a Control Group subject will NOT receive the Psychiatric Electroencephalogram Evaluation Registry (PEER) Interactive Report (of probable medication response) under investigation and will treat the Subject with Standard of Care. The subject will be blinded to group assignment and will provide the primary outcome measure - Quick Inventory of Depressive Symptomatology - Self Report 16 item questionnaire.
- Treatment (Active Comparator): Intervention - Psychiatric Electroencephalogram Evaluation Registry (PEER) Interactive Report - Treatment group subjects will undergo all procedures e.g. medication washout and baseline electroencephalogram, administered to the Control group. A clinician treating a Treatment Group subject will receive the Psychiatric Electroencephalogram Evaluation Registry (PEER) Report (of probable medication response) under investigation and will incorporate the Report information during prescription of medications to the Subject. The subject will be blinded to group assignment and will provide the primary outcome measure - Quick Inventory of Depressive Symptomatology - Self Report 16 item questionnaire.
  Interventions: Device: PEER Interactive Report

INTERVENTIONS:
Device: PEER Interactive Report — A subinvestigator treating a Treatment Group subject will receive the Psychiatric Electroencephalogram Evaluation Registry (PEER) Interactive Report (of probable medication response) under investigation and will incorporate the Report information during prescription of medications to the Subject. A subinvestigator treating a Control Group subject will NOT receive the PEER Report and will treat the Subject with Standard of Care. The subject will be blinded to group assignment and will provide the primary outcome measure - Quick Inventory of Depressive Symptomatology - Self Report 16 item questionnaire.
  Other Names: PEER Report
  Arms: Treatment

SUMMARY:
This is a prospective, multicenter, randomized, double-blind, controlled study to evaluate the effectiveness of Psychiatric Electroencephalogram Registry (PEER) Interactive to inform medication prescription in subjects with a primary diagnosis of depression with comorbidity of non-psychotic behavioral disorders versus treatment as usual, as determined by the investigator. The primary measurement for improvement of the subjects depression will be a self-evaluation questionnaire, the Quick Inventory of Depressive Symptomatology-Self Report 16 , but the investigators will also collect information on their clinical global improvement and any reduction in adverse events.

DETAILED DESCRIPTION:
This study is prospective in nature. Subjects in the control group will be treated according to treatment as usual and best judgment of the treating physician. For the experimental group the treating physician will follow the guidance of the subject's PEER Interactive Report as regards sensitivity to on-label medications and classes of medication.

The subjects will be washed out of all current medications prior to having an electroencephalogram (EEG), which is necessary to generate the PEER Interactive Report. The wash out period for outpatients is no longer than 14 days.

The subjects will be followed for 3 months after the initial treatment. The patient will be seen on a routine basis and assessments will be made at each interaction to evaluate the patient's improvement in mental health. The subjects will also be closely evaluated to determine if they are experiencing any psychiatric specific adverse events. The investigator is allowed to treat the patient according to their best medical judgment, which may include adding or changing medications, seeing the patient more frequently, or other interventions such as the use of sleep aids.

ELIGIBILITY:
Inclusion Criteria:

1. Male and female subjects between the ages of 18 - 65 years of age or older who speak and read English.
2. Subjects able to provide written informed consent to participate in the study.
3. Subjects with a primary diagnosis of a Diagnostic and Statistical Manual of Mental Disorders (DSM-V) depressive disorder. Please see Appendix D for definitions.
4. Subjects with comorbidity of a non-psychotic behavioral disorder. Please see Appendix D for definitions.
5. Subjects with comorbidity of mild traumatic brain injury (mTBI) are eligible for inclusion in this study.
6. Subjects with comorbidity of post-traumatic stress disorder (PTSD) are eligible for inclusion in this study. A score of 45 or greater on the PTSD Checklist Civilian (PCL-C) measurement tool will qualify a subject for inclusion of diagnosis of PTSD as a comorbid condition.
7. Able to stop specified medications, including drugs of abuse, for 5 half-lives of the medication(s). See Appendix E for a list of the withdrawal periods for medications. The potential subject's primary care physician may be consulted to make these determinations.
8. Able to be washed out of medications within 14 days, i.e. 5 half-lives are not longer than 14 days (See Appendix E).
9. Ability to comply with the requirements of the study.

   -

Exclusion Criteria:

1. Male and female subjects less than 18 years old or greater than 65 years old.
2. Subjects who cannot provide written informed consent.
3. Diagnosis of a psychotic disorder. Please see Appendix D for definitions.
4. History of, or current, open head brain trauma.
5. Subjects with comorbidity of traumatic brain injury (TBI) who experienced greater than 30 minutes loss of consciousness, greater than 24 hour alteration in consciousness or mental status, greater than 24 hours of post traumatic amnesia, or a Glasgow Coma Scale (best available score in first 24 hours) of less than 13.
6. Subjects who, in the opinion of the investigator would not be good candidates to be washed out of specified medications (Appendix E) and are unable to washout medications and/or supplements in a period of 14 days or less.
7. History of: craniotomy, cerebral metastases, cerebrovascular accident; current diagnosis of seizure disorder, schizophrenia, schizo-affective disorder, dementia, mental retardation, or major depression with psychotic features; or use of depot neuroleptics in last 12 months.
8. Clinically significant medical illness, including thyroid disorders, diabetes, etc., which cannot be remediated with medication, e.g. synthroid, insulin, etc.
9. Participation in any other therapeutic drug study within 60 days preceding inclusion.
10. Known pregnancy and/or lactation, or intent to become pregnant during this study.
11. Chronic or acute pain requiring prescription pain medication(s) (narcotic or synthetic narcotic).
12. Candidates with any metal, shrapnel or other similar objects in the head that could affect the QEEG.
13. Candidates currently stable on current medications.
14. Pre-entry subject whose urine drug screen is positive for drugs of abuse.

    -

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 468 (Estimated)
Dates: Start 2016-11; Primary Completion 2019-12 (Actual)

PRIMARY OUTCOMES:
Quick Inventory of Depressive Symptomatology - Self Report 16 questionnaire (QIDS-SR16) | 4 months
  A self reported survey - blinded subject acts as blinded rater/outcomes assessor. We will use this survey to measure the subject's self-reported change in symptoms of depression.

SECONDARY OUTCOMES:
Clinical Global Impressions - Improvement (CGI-I) | 4 months
  Commonly used measure of symptom severity, treatment response and the efficacy of treatments in treatment studies of patients with mental disorders
Clinical Global Impressions - Severity (CGI-S) | 4 months
  Commonly used measure of symptom severity, treatment response and the efficacy of treatments in treatment studies of patients with mental disorders.
Concise Health Risk Tracking Scale - 7 item Self Report Survey (CHRT- SR7) | 4 months
  A 7 question self-report questionnaire that assesses suicidal risk of subjects in clinical practice

CONTACTS AND LOCATIONS:
Overall Officials: Daniel Iosifescu, PhD, Principal Investigator — Mount Sinai Hospital, New York, N.Y.
Locations (1):
- Carolina Partners, Raleigh, North Carolina, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] DeBattista C, Kinrys G, Hoffman D, Goldstein C, Zajecka J, Kocsis J, Teicher M, Potkin S, Preda A, Multani G, Brandt L, Schiller M, Iosifescu D, Fava M. The use of referenced-EEG (rEEG) in assisting medication selection for the treatment of depression. J Psychiatr Res. 2011 Jan;45(1):64-75. doi: 10.1016/j.jpsychires.2010.05.009. Epub 2010 Jul 3. PMID 20598710
- [Background] Demyttenaere K, Desaiah D, Petit C, Croenlein J, Brecht S. Patient-assessed versus physician-assessed disease severity and outcome in patients with nonspecific pain associated with major depressive disorder. Prim Care Companion J Clin Psychiatry. 2009;11(1):8-15. doi: 10.4088/pcc.08m00670. PMID 19333404
- [Background] Duffy FH, Burchfiel JL, Lombroso CT. Brain electrical activity mapping (BEAM): a method for extending the clinical utility of EEG and evoked potential data. Ann Neurol. 1979 Apr;5(4):309-21. doi: 10.1002/ana.410050402. PMID 443765
- [Background] Hughes JR, John ER. Conventional and quantitative electroencephalography in psychiatry. J Neuropsychiatry Clin Neurosci. 1999 Spring;11(2):190-208. doi: 10.1176/jnp.11.2.190. PMID 10333991
- [Background] Hoffman DA, Debattista C, Valuck RJ, Iosifescu DV. Measuring severe adverse events and medication selection using a "PEER Report" for nonpsychotic patients: a retrospective chart review. Neuropsychiatr Dis Treat. 2012;8:277-84. doi: 10.2147/NDT.S31665. Epub 2012 Jun 21. PMID 22802691
- [Background] Rush AJ, Bernstein IH, Trivedi MH, Carmody TJ, Wisniewski S, Mundt JC, Shores-Wilson K, Biggs MM, Woo A, Nierenberg AA, Fava M. An evaluation of the quick inventory of depressive symptomatology and the hamilton rating scale for depression: a sequenced treatment alternatives to relieve depression trial report. Biol Psychiatry. 2006 Mar 15;59(6):493-501. doi: 10.1016/j.biopsych.2005.08.022. Epub 2005 Sep 30. PMID 16199008
- Available data/document: Study Protocol: CNSR012 Protocol — http://myndanalytics.com — Please email snavarre@myndanalytics.com for approved version of the protocol
- Available data/document: Informed Consent Form: CNSR012 ICD — http://myndanalytics.com — Please email snavarre@myndanalytics.com for approved version of ICD